CLINICAL TRIAL: NCT06482918
Title: Cognitive Remediation in Schizophrenia Patients: Study of the Efficacy and of the Role of Neuroplasticity in Two Different Approaches Based on "Top-down" and "Bottom-up" Mechanisms
Brief Title: Cognitive Remediation in Schizophrenia: Efficacy and Role of Neuroplasticity in "Top-down" and "Bottom-up" Mechanisms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, RODRIGO NIETO, MD PhD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fondecyt 11231216
Record Dates: First submitted 2024-06-19; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: Cognitive Remediation; Cognitive Training; Cognition; Brain-Derived Neurotrophic Factor
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Top-Down Cognitive Remediation (Experimental): Executive functions training
  Interventions: Behavioral: Cognitive Remediation
- Bottom-Up Cognitive Remediation (Experimental): Perceptual training
  Interventions: Behavioral: Cognitive Remediation
- Treatment-As-Usual (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive Remediation — Computer-assisted top-down or bottom-up cognitive remediation using tablets
  Arms: Bottom-Up Cognitive Remediation; Top-Down Cognitive Remediation

SUMMARY:
Schizophrenia patients have deficits of different degrees in several cognitive domains, impacting their social functioning and quality of life. Cognitive remediation strategies are useful to treat cognitive deficits in patients with schizophrenia. There are at least two different cognitive remediation strategies: one has a "top-down" approach, and is aimed at higher-order cognitive processes, focusing on the training of executive functions. The other one has a "bottom-up" approach, aiming to first recovering the perceptual processing alterations that may affect performance in higher-order cognitive functions. This study addresses in parallel two research questions, one of clinical interest (Are both strategies effective in improving neurocognitive performance?) and another one focused on the psychological / neurobiological mechanisms of neurocognitive remediation (Which cognitive remediation strategies are related to changes in BDNF levels?). The specific objectives are: (1) Evaluate the effectiveness of two cognitive remediation strategies. (2) Study the critical moments of neuroplasticity for each cognitive remediation strategy, observing changes in BDNF levels at the end of the intervention and 12 weeks after the intervention. (3) Identify potential clinical and/or molecular predictors (BDNF levels or val66met polymorphism) of response for each cognitive remediation strategy. For these objectives, two randomized controlled trials with two arms will be carried out in parallel, one where patients will receive cognitive remediation and another consisting of a control group (with usual treatment). The control group subjects will remain on a waiting and observation list for 10 weeks, to later enter the active arm, which will also last 10 weeks. In one of the trials the active arm will consist of cognitive remediation therapy with a "bottom-up" approach (focused on perceptual training), while in the other trial the active arm will consist of cognitive remediation with a "top-down" approach (focused on executive skills training). Neurocognitive and clinical assessments will be carried out along with the measurement of BDNF levels at four evaluation times: one at baseline, one at the end of the observation period with treatment-as-usual, another at the end of cognitive remediation, and another after a 12 week follow-up period.

DETAILED DESCRIPTION:
Schizophrenia is a severe psychiatric illness that has a significant impact on patients, their families, and society. It presents with deficits of different degrees in all cognitive domains, including memory, processing speed, attention and executive functions, which have been consistently demonstrated by different studies across several geographical regions. This has implications for patients' social functioning and quality of life, as cognitive symptoms together constitute the most important predictors of patients' functioning in the community. Antipsychotic drugs, although effective for psychotic symptoms, have little effect on cognition, however, cognitive rehabilitation achieves at least a medium effect size to improve cognition. There are at least two different cognitive remediation strategies, depending on the cognitive processes to which the intervention is targeted. One has a "top-down" approach, and is aimed at higher-order cognitive processes, and focuses on the training of executive functions. The other has a "bottom-up" approach and aims to first recovering the perceptual processing alterations that some patients with schizophrenia have and that would affect performance in higher-order cognitive functions.

This study addresses in parallel two research questions, one of clinical interest, and another focused on the psychological / neurobiological mechanisms of neurocognitive remediation: What neurocognitive remediation strategy, executive skills training ("top-down" approach) or training perceptual approach ("bottom-up" approach), is it effective in improving neurocognitive performance? Which neurocognitive remediation strategies are related to changes in BDNF levels? At what point of the recovery process are these changes observed? The hypothesis is that the "bottom-up" strategy presents observable results at the end of the intervention, whereas the "top-down" strategy results in an observable effect on neurocognitive performance and functioning in the community in a delayed manner, 12 weeks after the intervention. We expect that both strategies will be associated with an increase in BDNF levels compared to the situation prior to the intervention, but that this will occur at the time when the clinical effect is observed. The specific objectives are: (1) Evaluate the effectiveness of two cognitive remediation strategies, one focused on executive skills training (top-down approach) and another on perceptual training (bottom-up approach). (2) Study the critical moments of neuroplasticity for each cognitive remediation strategy, observing changes in BDNF levels at the end of the intervention and 12 weeks after the intervention. (3) Identify potential clinical and/or molecular predictors (BDNF levels or val66met polymorphism) of the response to treatment from the neurocognitive point of view for each cognitive remediation strategy.

In order to achieve this, two randomized controlled trials with two arms will be carried out in parallel, one where patients will receive cognitive remediation and another consisting of a control group (with usual treatment). The control group subjects will remain on a waiting and observation list for 10 weeks, to later enter the active arm, which will also last 10 weeks. In one of the trials the active arm will consist of cognitive remediation therapy with a "bottom-up" approach (focused on perceptual training), while in the other trial the active arm will consist of cognitive remediation with a "top-down" approach (focused on executive skills training). Neurocognitive and clinical assessments will be carried out along with the measurement of BDNF levels at four measurement times: one at baseline, one at the end of the observation period with treatment-as-usual, another at the end of cognitive remediation, and another after a 12 weeks follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to Diagnostic and Statistical Manual (DSM)-5
* Age between 18 and 59 years
* Clinically stable outpatients
* Current treatment with at least one antipsychotic medication

Exclusion Criteria:

* Significant medical or neurological comorbidity
* Substance use disorder with illegal drugs in active use
* Participation in a cognitive remediation program in the last 6 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
MCCB Global Cognition | After 10 weeks of cognitive remediation and at 12 week follow-up assessment
  Global Cognition Composite T Score in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
BDNF levels in peripheral blood | After 10 weeks of cognitive remediation and at 12 weeks follow-up assessment
  Brain-Derived Neurotrophic Factor levels in peripheral blood measured with ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo R. Nieto, MD PhD, Principal Investigator — University of Chile
Locations (1):
- Clinica Psiquiatrica Universitaria, Hospital Clinico de la Universidad de Chile, Santiago, RM, Chile

REFERENCES:
- [Background] Owen MJ, Sawa A, Mortensen PB. Schizophrenia. Lancet. 2016 Jul 2;388(10039):86-97. doi: 10.1016/S0140-6736(15)01121-6. Epub 2016 Jan 15. PMID 26777917
- [Background] Kahn RS, Sommer IE, Murray RM, Meyer-Lindenberg A, Weinberger DR, Cannon TD, O'Donovan M, Correll CU, Kane JM, van Os J, Insel TR. Schizophrenia. Nat Rev Dis Primers. 2015 Nov 12;1:15067. doi: 10.1038/nrdp.2015.67. PMID 27189524
- [Background] Schaefer J, Giangrande E, Weinberger DR, Dickinson D. The global cognitive impairment in schizophrenia: consistent over decades and around the world. Schizophr Res. 2013 Oct;150(1):42-50. doi: 10.1016/j.schres.2013.07.009. Epub 2013 Aug 2. PMID 23911259
- [Background] Green MF. What are the functional consequences of neurocognitive deficits in schizophrenia? Am J Psychiatry. 1996 Mar;153(3):321-30. doi: 10.1176/ajp.153.3.321. PMID 8610818
- [Background] Kuo SS, Almasy L, Gur RC, Prasad K, Roalf DR, Gur RE, Nimgaonkar VL, Pogue-Geile MF. Cognition and community functioning in schizophrenia: The nature of the relationship. J Abnorm Psychol. 2018 Feb;127(2):216-227. doi: 10.1037/abn0000326. PMID 29528675
- [Background] Keefe RS, Bilder RM, Davis SM, Harvey PD, Palmer BW, Gold JM, Meltzer HY, Green MF, Capuano G, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Davis CE, Hsiao JK, Lieberman JA; CATIE Investigators; Neurocognitive Working Group. Neurocognitive effects of antipsychotic medications in patients with chronic schizophrenia in the CATIE Trial. Arch Gen Psychiatry. 2007 Jun;64(6):633-47. doi: 10.1001/archpsyc.64.6.633. PMID 17548746
- [Background] Hori H, Noguchi H, Hashimoto R, Nakabayashi T, Omori M, Takahashi S, Tsukue R, Anami K, Hirabayashi N, Harada S, Saitoh O, Iwase M, Kajimoto O, Takeda M, Okabe S, Kunugi H. Antipsychotic medication and cognitive function in schizophrenia. Schizophr Res. 2006 Sep;86(1-3):138-46. doi: 10.1016/j.schres.2006.05.004. Epub 2006 Jun 21. PMID 16793238
- [Background] Moncrieff J, Cohen D, Mason JP. The subjective experience of taking antipsychotic medication: a content analysis of Internet data. Acta Psychiatr Scand. 2009 Aug;120(2):102-11. doi: 10.1111/j.1600-0447.2009.01356.x. Epub 2009 Feb 15. PMID 19222405
- [Background] McCleery A, Nuechterlein KH. Cognitive impairment in psychotic illness: prevalence, profile of impairment, developmental course, and treatment considerations . Dialogues Clin Neurosci. 2019 Sep;21(3):239-248. doi: 10.31887/DCNS.2019.21.3/amccleery. PMID 31749648
- [Background] Marder SR, Fenton W. Measurement and Treatment Research to Improve Cognition in Schizophrenia: NIMH MATRICS initiative to support the development of agents for improving cognition in schizophrenia. Schizophr Res. 2004 Dec 15;72(1):5-9. doi: 10.1016/j.schres.2004.09.010. PMID 15531402
- [Background] Green MF, Nuechterlein KH. The MATRICS initiative: developing a consensus cognitive battery for clinical trials. Schizophr Res. 2004 Dec 15;72(1):1-3. doi: 10.1016/j.schres.2004.09.006. No abstract available. PMID 15531401
- [Background] Best MW, Milanovic M, Iftene F, Bowie CR. A Randomized Controlled Trial of Executive Functioning Training Compared With Perceptual Training for Schizophrenia Spectrum Disorders: Effects on Neurophysiology, Neurocognition, and Functioning. Am J Psychiatry. 2019 Apr 1;176(4):297-306. doi: 10.1176/appi.ajp.2018.18070849. Epub 2019 Mar 8. PMID 30845819
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233
- [Background] Wykes T, Huddy V, Cellard C, McGurk SR, Czobor P. A meta-analysis of cognitive remediation for schizophrenia: methodology and effect sizes. Am J Psychiatry. 2011 May;168(5):472-85. doi: 10.1176/appi.ajp.2010.10060855. Epub 2011 Mar 15. PMID 21406461
- [Background] Lejeune JA, Northrop A, Kurtz MM. A Meta-analysis of Cognitive Remediation for Schizophrenia: Efficacy and the Role of Participant and Treatment Factors. Schizophr Bull. 2021 Jul 8;47(4):997-1006. doi: 10.1093/schbul/sbab022. PMID 33772310
- [Background] Vita A, Barlati S, Ceraso A, Nibbio G, Ariu C, Deste G, Wykes T. Effectiveness, Core Elements, and Moderators of Response of Cognitive Remediation for Schizophrenia: A Systematic Review and Meta-analysis of Randomized Clinical Trials. JAMA Psychiatry. 2021 Aug 1;78(8):848-858. doi: 10.1001/jamapsychiatry.2021.0620. PMID 33877289
- [Background] Adcock RA, Dale C, Fisher M, Aldebot S, Genevsky A, Simpson GV, Nagarajan S, Vinogradov S. When top-down meets bottom-up: auditory training enhances verbal memory in schizophrenia. Schizophr Bull. 2009 Nov;35(6):1132-41. doi: 10.1093/schbul/sbp068. Epub 2009 Sep 10. PMID 19745022
- [Background] Vinogradov S. Has the Time Come for Cognitive Remediation in Schizophrenia...Again? Am J Psychiatry. 2019 Apr 1;176(4):262-264. doi: 10.1176/appi.ajp.2019.19020160. No abstract available. PMID 30929502